CLINICAL TRIAL: NCT03298893
Title: A Phase-I Study of Nivolumab in Association With Radiotherapy and Cisplatin in Locally Advanced Cervical Cancers Followed by Adjuvant Nivolumab for up to 6 Months. NiCOL
Brief Title: Nivolumab in Association With Radiotherapy and Cisplatin in Locally Advanced Cervical Cancers Followed by Adjuvant Nivolumab for up to 6 Months (NiCOL)
Acronym: NiCOL
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Institut Curie (Other)
Collaborators: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IC 2016-08
Record Dates: First submitted 2017-09-27; First posted 2017-10-02 (Actual); Last update posted 2025-09-19 (Actual); Status verified 2025-09

CONDITIONS: Cervical Cancer; Locally Advanced Cervical Cancer
Keywords: cervical cancer; nivolumab; cisplatin; radiotherapy
MeSH Terms: conditions — Uterine Cervical Neoplasms | interventions — Nivolumab; Cisplatin; Radiotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Nivolumab + radiochemotherapy (Experimental): 5 weeks of radiochemotherapy + nivolumab followed by 5 months of nivolumab alone
  Interventions: Drug: Nivolumab Injection; Drug: Cisplatin; Radiation: radiotherapy

INTERVENTIONS:
Drug: Nivolumab Injection — 2 possible doses : flat dose 240 mg q2 weeks or 1mg/kg q2 weeks
Drug: Cisplatin — 40 mg/m2, once a week during radiotherapy
Radiation: radiotherapy — Intensity-modulated radiation therapy (including volumetric-modulated arc therapy and tomography) will be used. A dose of 45 Gy will be delivered to the pelvis in 25 fractions of 1.8 Gy using a 6-MV photon energy.
  An additional dose of 54 Gy in 25 fractions of 2.16 Gy may be delivered to invaded lymph nodes using SIB-IMRT.
  An additional lateral pelvic dose may be delivered if coverage of the target volumes is judged insufficient. The volumes, doses and techniques will be those usually used in each center.

SUMMARY:
To date, the majority of clinical trials on checkpoint inhibitors have tested these agents as monotherapy, and the next logical step is to evaluate rational therapeutic associations. The aim of the NiCOL study is to assess the safety of nivolumab in association with chemoradiation therapy and to gain initial insight into its efficacy in association with the current standard of care, including chemoradiation.

ELIGIBILITY:
Inclusion Criteria:

1. Adult patients at least 18 years of age;
2. Ability to understand and the willingness to sign a written informed consent document.;
3. Eastern Cooperative Oncology Group (ECOG) Performance Status 0 or 1;
4. Histologically confirmed locally advanced cervical cancer, i.e. FIGO stages IB2 to IVA, squamous-cell carcinoma or adenocarcinoma, with indication for radiotherapy and cisplatin-based chemotherapy with a curative intent as confirmed by a multidisciplinary board including a radiation oncologist. PD-L1 expression on tumor will not be required for inclusion; (staging may include [18F]-fluorodeoxyglucose (FDG) PET-CT and/or para-aortic dissection in accordance with usual practice in each investigational center and at the Investigator's discretion);
5. Disease amenable to biopsy since three tumor samples are mandatory prior to treatment;
6. Laboratory values at Screening must meet the following criteria :

   neutrophils ≥ 1.0 x 109/L, lymphocytes ≥ 0.5 x 109/L, platelets ≥ 100 x 109/L, hemoglobin ≥ 8.0 g/dL, creatinine ≤ 2 times the upper limit of normal (ULN), aspartate aminotransferase (AST) ≤ 3 ULN, alanine aminotransferase (ALT) ≤ 3 x ULN, total bilirubin ≤ 1.5 x ULN (≤ 3 x ULN if genetically documented Gilbert's syndrome).
7. For women with child-bearing potential, negative blood or urinary pregnancy test within 24 hours of initiation of nivolumab, as well as appropriate method of contraception throughout the study ;
8. Affiliated to the French Social Security System.

Exclusion Criteria:

1. Metastases (except pelvic and/or para-aortic nodal metastases) ;
2. Peritoneal carcinosis;
3. Sensory or motor neuropathy ≥ grade 2;
4. Active or recent history of known autoimmune disease or recent history of a syndrome that required systemic corticosteroids or immunosuppressive drugs, except for :

   * hydrocortisone, which is permitted at physiological doses;
   * syndromes that would not be expected to recur in the absence of an external trigger, e.g. glomerulonephritis;
   * vitiligo or autoimmune thyroiditis;
5. Type-1 or type-2 diabetes;
6. History of or current immunodeficiency disease, including known history of infection with human immunodeficiency virus;
7. Prior systemic treatment or radiotherapy for cervical cancer;
8. Prior allogeneic stem cell transplantation;
9. Prior immunotherapy, including tumor vaccine, cytokine, anti-CTLA4, anti-PD-1, anti-PD-L1 or similar agents;
10. Any non-oncologic vaccine for prevention of infectious disease within 28 days prior to inclusion, including but not limited to measles, mumps, rubella, chicken pox, yellow fever, seasonal influenza, H1N1, rabies, BCG, and typhoid vaccine;
11. Positive serology for hepatitis B surface antigen;
12. Positive for hepatitis-C ribonucleic acid on polymerase chain reaction;
13. Active infection requiring therapy;
14. History of idiopathic pulmonary fibrosis (including pneumonitis), drug-induced pneumonitis, organizing pneumonia or evidence of active pneumonitis on chest CT-scan at Screening;
15. History of malignancy (excepting non-melanoma skin cancer) unless complete remission was achieved at least 3 years prior to inclusion and no additional therapy is required or planned during the study;
16. Underlying medical condition that, in the Investigator's opinion, could render the administration of the study treatment hazardous; additional severe and/or uncontrolled concurrent disease;
17. Concomitant use of other investigational drugs;
18. Pregnancy or breastfeeding.

Ages: 18 Years to 99 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2017-11-27 (Actual); Primary Completion 2020-10-30 (Actual); Study Completion 2022-03-07 (Actual)

PRIMARY OUTCOMES:
rate of occurrence of dose-limiting toxicity (DLT) | within 11 weeks after the initiation of treatment.
  DLT is defined as any of the following treatment-related adverse events or laboratory abnormalities, graded according to National Cancer Institute Common Terminology Criteria for Adverse Events (NCI-CTCAE) version 4.0:
  * non-hematological toxicity ≥ grade 3;
  * immune-related adverse event ≥ grade 3;
  * symptomatic immune-related adverse event ≥ grade 2 resistant to optimal supportive care for > 7 days;
  * dosing delay in RT ≥ 1 week due to toxicity related to nivolumab, chemotherapy or RT;
  * colitis or diarrhea ≥ grade 3.

SECONDARY OUTCOMES:
Objective Response Rate (ORR) | after the end of RT and before brachytherapy and again up to 2 months after brachytherapy
  ORR is defined as the proportion of all subjects whose best response is either a complete response or a partial response.
Progression Free Survival (PFS) | 2 years
  PFS is defined as the length of time from the start of treatment to disease progression or death, regardless of the cause of death
Disease Free Survival (DFS) | 2 years
  DFS is defined as the length of time from the start of complete response to the time of relapse from complete response. DFS applies only to patients in complete response.
Incidence of Serious Adverse Events (SAEs) to assess the overall safety profile of the association of nivolumab and pelvic radio-chemotherapy | from the first intake of the IMP until 100 days after the last intake of the IMP
Incidence of Adverse Events (AEs) to assess the overall safety profile of the association of nivolumab and pelvic radio-chemotherapy | from the first intake of the IMP until 100 days after the last intake of the IMP
validation of molecular alterations detected by molecular analyses | 2 years
  Retrospective exome, RNA and targeted sequencing analyses will be performed on all patients treated and for whom tumor samples are available.
ctDNA heterogeneity | baseline, at Weeks 3, 6 and 12 and every 12 weeks up to Week 104
  Retrospective exome and targeted sequencing analyses will be performed on all patients treated and for whom tissue samples are available at the different timepoints
tumor microenvironment description | 2 years
  phenotypic analysis of the different components of the tumor microenvironment using various technologies
tumor PD-L1 immunohistochemistry | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Emanuela Romano, MD, Study Director — Institut Curie
Locations (3):
- France (3):
  - Institut Curie, Paris
  - Hopital Européen Georges Pompidou, Paris
  - Institut Curie Hopital René Huguenin, Saint-Cloud

IPD SHARING:
Plan to Share IPD: Yes
Sponsor will share de-identified data sets. Documents generated under the project will be disseminated in accordance with Institut Curie policies.
Supporting Information: Study Protocol, SAP
Time Frame: Data requests can be submitted starting 9 months after last article publication and will be made accessible for up to 12 months.
Access Criteria: Access to trial individual participant data can be requested by qualified researchers engaging in independent scientific research, and will be provided following review and approval of a research proposal and Statistical Analysis Plan (SAP) and execution of a data sharing agreement (DSA).

REFERENCES:
- [Result] Rodrigues M, Vanoni G, Loap P, Dubot C, Timperi E, Minsat M, Bazire L, Durdux C, Fourchotte V, Laas E, Pouget N, Castel-Ajgal Z, Marret G, Lesage L, Meseure D, Vincent-Salomon A, Lecompte L, Servant N, Vacher S, Bieche I, Malhaire C, Huchet V, Champion L, Kamal M, Amigorena S, Lantz O, Chevrier M, Romano E. Nivolumab plus chemoradiotherapy in locally-advanced cervical cancer: the NICOL phase 1 trial. Nat Commun. 2023 Jun 22;14(1):3698. doi: 10.1038/s41467-023-39383-8. PMID 37349318